CLINICAL TRIAL: NCT03959202
Title: A Personalized Behavioral Intervention to Improve Physical Activity, Sleep and Cognition in Sedentary Older Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00198497; R00NR016484 (NIH)
Record Dates: First submitted 2019-05-20; First posted 2019-05-22 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2022-07

CONDITIONS: Sleep
Keywords: older adults; exercise intervention; cognition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Based on the self-efficacy theory, participants in the intervention arm will receive personalized, circadian-based activity guidelines, a 2-hour in person education session, real time physical activity self-monitoring, interactive prompts, biweekly phone consultation with the research team, and financial incentives for achieving weekly physical activity goal.
  Interventions: Behavioral: ELDERFITNESS
- Control (Placebo Comparator): The control group will receive general education on physical activity for older adults and continue daily activity and healthcare routine. Participants in this group will also receive a Go4Life program book from the National Institute on Aging.
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: ELDERFITNESS — In-person training with the exercise trainer ( 3 sessions for participants without cognitive impairments over 24 weeks & 4 sessions for older adults with mild cognitive impairment over 16 weeks). Self-monitoring level of physical activity (steps & minutes of moderate activity) using the smart watch. . The Google calendar and Fitbit apps will send messages and alerts to the subject's smart watch that encourage subjects to achieve subjects' daily goals. If a participant has low activity for 3 consecutive days, the research assistant will call the participant to either encourage the participant to adhere to the plan or provide a modified plan after consulting the exercise trainer. Phone consultation: Subjects will have biweekly phone consultation with the research team members to receive guidance and adjustment on activity plans.Financial incentives: when the daily activity goal is achieved for more than four days per week, a $5 reward will be given to subjects.
  Arms: Intervention
Other: Control — General Education on physical activity for older adults and continue daily activity and healthcare routine. Participants will also receive a Go4Life Program book from the National Institute on Aging
  Arms: Control

SUMMARY:
Cognitive decline and sleep complaints are prevalent in older adults and severely affect older adults' physical health and quality of life. Sedentary lifestyle, which is reported by 90% of older Americans, is an important risk factor for both cognitive decline and sleep disturbances. Although promoting physical activity has benefits to older adults' health, including sleep and cognition, traditional interventions to increase activity are challenging due to extensive staffing requirements and low adherence. Electronic activity monitors, such as wrist-worn accelerometers, can track heart rate, activity, and sleep to allow individuals to work towards personal activity and sleep goals. These appealing features make these devices ideal for interventions that aim to change behaviors and improve health outcomes. However, the efficacy of using electronic activity monitors to promote physical activity and health in older adults has not been examined.

The investigators will conduct a randomized controlled trial in a cohort of older adults (without dementia) with both sedentary lifestyle and nocturnal sleep complaints to examine the effectiveness of a personalized behavioral intervention (compared to a control group) embedded within a smart watch application in older adults. 94 cognitively intact elders and 21 older adults with mild cognitive impairment will be enrolled and randomly allocated to the intervention or control group. Participants in the intervention arm will receive in person exercise training sessions, and personalized, self-monitor physical activity, receive interactive prompts, biweekly phone consultation with the research team, and financial incentives for achieving weekly physical activity goals. The control group will receive general education on physical activity in older adults and continue the routine daily activity during the intervention period. The intervention for older adults without cognitive impairment is 24 weeks and for older adults with mild cognitive impairment is 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Intact cognition or mild cognitive impairment
* Poor sleep quality
* Approval from healthcare provider to engage in mild to moderate physical activity
* More than 5 hours of self-reported sedentary time per day
* Understands English

Exclusion Criteria:

* Untreated sleep apnea as diagnosed by polysomnography

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2019-07-11 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Change in Objective Sleep Duration | Week 1, Week 26 intact cognition or Week 18 for mild cognitive impairment (MCI)
  Total Sleep time (minutes) will be measured using actigraph
Change in Sleep Efficiency as Assessed by Actigraphy | Week 1, Week 26 intact cognition or Week 18 for MCI
  Sleep efficiency (reported as a percentage) will be measured using actigraphy
Change in Subjective Sleep Quality as Assessed by the Pittsburgh Sleep Quality Index (PSQI) | Week 1, Week 26 intact cognition or Week 18 for MCI
  The PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Change in Plasma tumor necrosis factor-α (TNF-α) | Week 1, Week 26 intact cognition or Week 18 for MCI
  The TNF (pg/mL) will be measured using Plasma from blood draw
Change in Plasma C-reactive protein (CRP) | Week 1, Week 26 intact cognition or Week 18 for MCI
  The CRP (pg/mL) will be measured using Plasma from blood draw
Change in Plasma interleukin-6 (IL-6) | Week 1, Week 26 intact cognition or Week 18 for MCI
  The IL-6 (pg/mL) will be measured using Plasma from blood draw
Change in Plasma interleukin-1ß (IL-1ß) | Week 1, Week 26 intact cognition or Week 18 for MCI
  The IL-1ß (pg/mL) will be measured using Plasma from blood draw
Change in Global Cognition As Assessed by The Cogstate Brief Battery (CBB) | Week 1, Week 26 intact cognition or Week 18 for MCI
  The Cogstate Brief Battery (CBB) will be used as the primary assessment of cognitive function. The CBB is a computer based cognitive battery that scores four core cognitive domains: processing speed, attention/vigilance, visual learning memory and visual working memory. The composite cognition score is the primary cognition measure used to measure global cognitive function. The score will range from 0-400, with a higher score indicating higher performance.
Change in Physical Activity (PA) as Assessed by Actigraphy | Week 1, Week 26 intact cognition or Week 18 for MCI
  The Actigraphy (counts/min) will be used as a standardized research tool for PA assessment. Higher counts/min indicate higher level of physical activity.
Change in Physical Activity (PA) as assessed by the Physical Activity Scale for the Elderly | Week 1, Week 26 intact cognition or Week 18 for MCI
  Subjective PA will be obtained from the Physical Activity Scale for the Elderly. Score ranges from 0-400. The higher the score the higher the physical activity level.

CONTACTS AND LOCATIONS:
Overall Officials: Junxin Li, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No